CLINICAL TRIAL: NCT06382363
Title: Improving T2DM Detection Among At-Risk Individuals - Effectiveness of Active Opportunistic Screening Using Spot Capillary-HbA1c Test - a Cluster Randomized Controlled Trial (DM-REACH)
Brief Title: Improving T2DM Detection Using Spot cHbA1c Test
Acronym: DM-REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government); Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Linda Chan, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UW21-363
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus; Pre-diabetes
Keywords: Hemoglobin-A1c; Screening; Point-of-Care Testing
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects in the control group will be offered a free venous HbA1c test. Consistent with current practice at GOPCs, the venous sampling will be scheduled on a separate clinic visit at a set time within 1-2 weeks of recruitment. Test results will be available within one week. The subject will be informed via phone call regarding his/her DM risk, and if his/her HbA1c≥5.6%, he/she will be scheduled for a confirmatory OGTT within 2-4 weeks, ideally at the same clinic.
- Intervention (Experimental): Subjects in the intervention group will be offered a free POC-cHbA1c test to screen for hyperglycemia. The test will be performed on-site (i.e. during the same clinic visit of recruitment). Test results will be available within 10 minutes and the subject will be immediately informed of his/her DM risk, and for those with HbA1c≥5.6%, a confirmatory OGTT will be arranged on-site, scheduled within 2-4 weeks and ideally at the same clinic.
  Interventions: Procedure: POC-cHbA1c testing

INTERVENTIONS:
Procedure: POC-cHbA1c testing — The point-of-care HbA1c instrument employed in this study will be the Cobas b 101 (Roche Diagnostics, Switzerland) diagnostic test system. A capillary blood sample will be obtained by dermal puncture of a fingertip using a disposable lancet and resorbed in the specially marked area of the Cobas b 101 test disc. The disc will be inserted in the autoanalyzer. Test results displayed in both % and mmol/l will be available within 10 minutes.
  Arms: Intervention

SUMMARY:
Objectives: To evaluate the effectiveness of active opportunistic screening using point-of-care capillary Hemoglobin-A1c (POC-cHbA1c) testing, compared to venous HbA1c (vHbA1c) testing, in improving detection of type 2 diabetes mellitus (T2DM) among at-risk primary care patients.

Design: Pragmatic cluster randomized controlled trial.

Setting: 8 public primary care clinics in Hong Kong.

Participants: A minimum of 776 patients (97 per clinic) who have ≥1 risk factor for T2DM, but no known diagnosis of DM or DM screening in the past 12 months.

Intervention: Participants at intervention clinics (n=4) will be offered free POC-cHbA1c testing on-site, immediately informed of test results and DM risk, and scheduled for confirmatory oral glucose tolerance test (OGTT) if screened positive (i.e. HbA1c≥5.6%). Participants at control clinics will be offered free vHbA1c testing scheduled on a separate day, informed of test results and DM risk via phone, and scheduled for confirmatory OGTT if screened positive.

Main outcome measures: Primary outcomes are uptake rate of POC-cHbA1c versus vHba1c testing, and difference in proportion of T2DM detected between intervention and control groups.

Secondary outcomes include number-needed-to-screen to detect one more T2DM case.

Data analysis: Participants' characteristics and test uptake rates will be summarized by descriptive statistics. Difference in the proportion of T2DM detected between groups will be compared using Chi-squared test. Number-needed-to screen to identify one additional patient with DM will be calculated.

Expected results: A greater proportion of T2DM patients will be detected by POC-cHbA1c than vHbA1c due to a higher screening test uptake rate among the studied population.

DETAILED DESCRIPTION:
Aim:

This pragmatic cluster randomized controlled trial aims to determine the effectiveness of active opportunistic screening using point-of-care capillary HbA1c (POC-cHbA1c) testing compared to venous HbA1c (vHbA1c) testing in improving T2DM detection among at-risk public primary care patients, to estimate the impact of such a screening strategy in the real-world setting. The ultimate goal would be to fill the current preventive care gap and reduce the burden of undiagnosed T2DM in Hong Kong.

Objectives:

Primary Objectives

1. To determine the difference in the proportion of T2DM detected between the intervention group (POC-cHbA1c testing) and control group (conventional vHbA1c testing).
2. To evaluate the uptake rate of the POC-cHbA1c test relative to the vHbA1c test among at-risk public primary care patients in Hong Kong.

Secondary Objectives

1. To determine the proportion of subjects with high-risk HbA1c concentration (i.e. HbA1c≥5.6%) among the studied at-risk group.
2. To compare the difference in uptake rate of confirmatory OGTT test between intervention and control groups.
3. To calculate the number-needed-to-screen to detect one more case with T2DM using POC-cHbA1c testing compared to vHbA1c testing.
4. The proportion of patients who refuse to join the study (among all eligible subjects).

Hypotheses:

1. A greater proportion of T2DM patients will be detected in the intervention group (POC-cHbA1c testing) than in the control group (vHbA1c).
2. Uptake rate of POC-cHbA1c testing will be higher than vHbA1c testing among the studied population.
3. Uptake rate of confirmatory OGTT among screened positive patients (i.e. HbA1c ≥5.6%) in the intervention group will be higher than for those in the control group.

Data analysis:

Descriptive statistics will be used to summarize patients' characteristics in the intervention (POC-cHbA1c testing) group and control (vHbA1c testing) group. The difference in characteristics between groups will be assessed by independent t-tests for continuous variables or Chi-square tests for categorical variables. The uptake rate of POC-cHbA1c testing and vHbA1c testing will be reported. The difference in the proportion of T2DM detected between groups will also be compared using a Chi-squared test. The number-needed-to-screen to identify one additional patient with DM will be calculated. To take cluster effect into account, a mixed effect logistic model will be used to evaluate the effect of the intervention on the uptake rate by treating the clinic as a random effect and adjusting for the patients' characteristics. All statistical analyses will be performed using Stata. All significance tests will be two-tailed and findings with a p-value less than 0.05 will be considered statistically significant.

Potential problem:

Missing data will be handled by using multiple imputation. The chained equation method will be used to impute each missing value five times, adjusted for all baseline covariates and outcomes. The same analysis method will be adopted for each of the five imputed datasets, and the results will be pooled using Rubin's rule. Complete case analysis will also be conducted to confirm the results by multiple imputation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic patient;
* Aged ≥ 45 years;
* Family history of DM in a first-degree relative;
* History of Gestational DM;
* Hypertension (i.e. Systolic Blood Pressure (BP) ≥140mmHg, Diastolic BP ≥90mmHg or on therapy for hypertension);
* History of pre-diabetes (i.e. impaired fasting glucose with fasting glucose concentration between 5.6-6.9 mmol/L, impaired glucose tolerance with 2-hour post challenge plasma glucose concentration between 7.8-11.0 mmol/L or HbA1c between 5.6-6.4%);
* Hyperlipidemia (i.e. total cholesterol ≥ 5.2 mmol/L, triglycerides ≥ 1.7 mmol/L or on therapy);
* Obesity (i.e. for Chinese subjects, body mass index (BMI) ≥ 25 kg/m2).

Exclusion Criteria:

* Known history of T2DM or on hypoglycaemic treatment;
* Received T2DM screening within 12-months;
* Women who are pregnant or breast-feeding at recruitment;
* Active thyroid diseases (including subjects on thyroid replacement therapy or anti-thyroid drugs) or active endocrine diseases such as Cushing's syndrome or Acromegaly at recruitment;
* History of blood donation or blood transfusion within 3 months prior to recruitment;
* Patients who are taking systemic steroid therapy or iron supplement at recruitment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2022-06-11 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Proportional difference in detection of T2DM | 36 months
  The difference in proportion of T2DM detected between the intervention group (POC-cHbA1c testing) and control group (vHbA1c testing)
Uptake rate | 36 months
  The uptake rate of POC-cHbA1c testing and vHbA1c testing among consented participants

SECONDARY OUTCOMES:
Proportion of high-risk HbA1c concentration | 36 months
  The proportion of subjects with high-risk HbA1c concentration ≥5.6% among the studied at-risk group
Difference in uptake rate of OGTT | 36 months
  The difference in the uptake rate of confirmatory OGTT between intervention and control groups
Number-needed-to-screen to detect one more T2DM case | 36 months
  The number-needed-to-screen for POC-cHbA1c to detect one more case with T2DM compared to vHbA1c testing
Proportion of patients who refuse to join the study | 36 months
  The proportion of patients who refuse to join the study (among all eligible subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Chan, Principal Investigator — The University of Hong Kong
Locations (8):
- Hong Kong (8):
  - Aberdeen Jockey Club General Out-Patient Clinic, Hong Kong
  - Kwun Tong Community Health Centre, Hong Kong
  - Lek Yuen General Out-Patient Clinic, Hong Kong
  - Li Po Chun General Out-Patient Clinic, Hong Kong
  - Ma On Shan Family Medicine Centre, Hong Kong
  - Sai Ying Pun Jockey Club General Out-patient Clinic, Hong Kong
  - Tseung Kwan O (Po Ning Road) General Out-patient Clinic, Hong Kong
  - Yau Ma Tei Jockey Club Specialist Clinic, Hong Kong

REFERENCES:
- [Derived] Chan L, Yu EYT, Wan EYF, Wong SYS, Chao DVK, Ko WWK, Chen CXR, Chan PPL, Bilney EVM, Lee ES, Ng WL, Lam CLK. Improving type 2 diabetes detection among at-risk individuals - comparing the effectiveness of active opportunistic screening using spot capillary-HbA1c testing and venous HbA1c testing: a cluster randomized controlled trial. BMC Med. 2025 Mar 31;23(1):190. doi: 10.1186/s12916-025-04007-z. PMID 40165254